CLINICAL TRIAL: NCT00136357
Title: Treatment of Posttraumatic Stress Disorder in Kosovar High School Students Using Mind-Body Skills Groups: A Randomized Controlled Trial
Brief Title: Treatment of Posttraumatic Stress Disorder in Kosovar High School Students Using Mind-Body Skills Groups
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Center for Mind-Body Medicine (Other)
Responsible Party: Principal Investigator, James S. Gordon, M.D., Founder and Director, The Center for Mind-Body Medicine
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: MBSG 2004-01
Record Dates: First submitted 2005-08-26; First posted 2005-08-29 (Estimated); Results first posted 2015-02-16 (Estimated); Last update posted 2015-02-16 (Estimated); Status verified 2015-02

CONDITIONS: Stress Disorders, Post-traumatic
Keywords: posttraumatic stress; mind-body techniques; war; adolescents
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Mind-Body Skills Groups (Experimental): 12 week mind-body skills group program including guided imagery, relaxation techniques,autogenic training, meditation, biofeedback, drawings, genograms and movement techniques.
  Interventions: Behavioral: Mind-Body Skills Groups
- Delayed Intervention (No Intervention): Comparison group not receiving intervention until after the initial intervention was completed.

INTERVENTIONS:
Behavioral: Mind-Body Skills Groups — 12 week mind-body skills group program including guided imagery, relaxation techniques,autogenic training, meditation, biofeedback, drawings, genograms and movement techniques.
  Arms: Mind-Body Skills Groups

SUMMARY:
The purpose of this study is to determine whether the participation in a group program which includes meditation, biofeedback, drawings, autogenic training, genograms, and a variety of movement and breathing techniques will decrease symptoms of posttraumatic stress in high school students.

DETAILED DESCRIPTION:
The objective of this study is to determine whether participation in a group program incorporating mind-body techniques decreases symptoms of posttraumatic stress in adolescents. Students will be screened for posttraumatic stress using the Harvard Trauma Questionnaire and eighty-two qualifying students will be randomly assigned to a 12-session mind-body group program or a wait-list delayed intervention group. The program will be conducted by the teachers at a high school in Kosovo and include meditation, biofeedback, drawings, autogenic training, genograms, and a variety of movement and breathing techniques. Changes in posttraumatic stress symptoms will be measured using the Harvard Trauma Questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Students having posttraumatic stress (PTSD) as defined according to a scoring algorithm of the Harvard Trauma Questionnaire previously described by the Harvard Refugee Trauma group and used in a Kosovar Albanian population. This definition of PTSD requires a score of 3 or 4, on a Likert scale of 1-4, on at least one of the four of the reexperiencing symptoms (Criterion B), at least 3 of the 7 avoidance and numbing symptoms (Criterion C), and at least 2 of the 5 arousal symptoms (Criterion D) in addition to exposure to a traumatic event (Criterion A).

Exclusion Criteria:

* No specific exclusion criteria. Students having PTSD symptoms as defined above may participate in the study.

Ages: 14 Years to 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 82 (Actual)
Dates: Start 2004-08; Primary Completion 2005-05 (Actual); Study Completion 2005-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James S Gordon, MD, Principal Investigator — The Center for Mind-Body Medicine
Locations (1):
- Jeta e Re High School, Suhareka, Kosovo, Federal Republic of Yugoslavia

REFERENCES:
- [Background] Gordon JS, Staples JK, Blyta A, Bytyqi M. Treatment of posttraumatic stress disorder in postwar Kosovo high school students using mind-body skills groups: a pilot study. J Trauma Stress. 2004 Apr;17(2):143-7. doi: 10.1023/B:JOTS.0000022620.13209.a0. PMID 15141787
- [Derived] Gordon JS, Staples JK, Blyta A, Bytyqi M, Wilson AT. Treatment of posttraumatic stress disorder in postwar Kosovar adolescents using mind-body skills groups: a randomized controlled trial. J Clin Psychiatry. 2008 Sep;69(9):1469-76. doi: 10.4088/jcp.v69n0915. Epub 2008 Aug 1. PMID 18945398
- See also: Center for Mind-Body Medicine website — http://www.cmbm.org

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Mind-Body Skills Groups | Delayed Intervention
Started | 41 | 41
Completed | 38 | 39
Not Completed | 3 | 2
Not completed — Withdrawal by Subject | 3 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Mind-Body Skills Groups | Delayed Intervention | Total
Number analyzed (Participants) | 41 | 41 | 82
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 41 | 41 | 82
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 16.3 (1.1) | 16.3 (1.2) | 16.3 (1.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31 | 31 | 62
  Male | 10 | 10 | 20
Region of Enrollment [Number; unit: participants]
  Kosovo | 41 | 41 | 82

OUTCOME MEASURES:

1. Primary Outcome: Harvard Trauma Questionnaire
Description: The Harvard Trauma Questionnaire measures PTSD Symptoms. This scale has 16 items and is rated on a Likert scale from 1-4. The total score is sum of the scores divided by the number of items. Higher scores indicated higher levels of PTSD symptoms.
Time Frame: Baseline, 12 weeks, 3 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Mind-Body Skills Groups | Delayed Intervention
Number analyzed (Participants) | 38 | 39
units on a scale
  Baseline | 2.5 (0.3) | 2.5 (0.3)
  12 Week Assessment | 2.0 (0.3) | 2.4 (0.4)
  3 Month Assessment | 2.0 (0.3) | 2.1 (0.3)

ADVERSE EVENTS:
Arm/Group | Mind-Body Skills Groups | Delayed Intervention
Serious Adverse Events (participants affected / at risk) | 0/41 | 0/41
Other Adverse Events (participants affected / at risk) | 0/41 | 0/41

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes